CLINICAL TRIAL: NCT01356888
Title: BIOTRONIK-Safety and Clinical PerFormance of the Drug ELuting Orsiro Stent in the Treatment of Subjects With Single de Novo Coronary Artery Lesions - II
Brief Title: Study of the Orsiro Drug Eluting Stent System
Acronym: BIOFLOW-II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C1004
Record Dates: First submitted 2011-05-18; First posted 2011-05-20 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Abbott Laboratories - Xience Prime DES (Active Comparator)
  Interventions: Device: Percutaneous Coronary Intervention (Abbott Laboratories - Xience Prime DES)
- Biotronik - Orsiro DES (Experimental)
  Interventions: Device: Percutaneous Coronary Intervention (Orsiro DES)

INTERVENTIONS:
Device: Percutaneous Coronary Intervention (Abbott Laboratories - Xience Prime DES) — Stenting
  Arms: Abbott Laboratories - Xience Prime DES
Device: Percutaneous Coronary Intervention (Orsiro DES) — stenting
  Arms: Biotronik - Orsiro DES

SUMMARY:
The purpose of this study is to compare the BIOTRONIK Orsiro Drug Eluting Stent System with the Abbott Xience Prime™ Drug Eluting Stent System with respect to in-stent Late Lumen Loss in a non-inferiority study in de novo coronary lesions at 9 months.

ELIGIBILITY:
Main Inclusion Criteria:

* Subject has provided a written informed consent
* Single de novo lesion with ≥ 50% and <100% stenosis in up to 2 coronary arteries
* The target lesion length is ≤ 26 mm
* The target reference vessel diameter is ≥ 2.25 mm and ≤ 4.0 mm

Main Exclusion Criteria:

* Evidence of myocardial infarction within 72 hours prior to index procedure
* Unprotected left main coronary artery disease (stenosis >50%)
* Three-vessel coronary artery disease at time of procedure Thrombus in target vessel
* Target lesion involves a side branch > 2.0 mm in diameter
* Heavily calcified lesion
* Target lesion is located in or supplied by an arterial or venous bypass graft

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2011-05; Primary Completion 2013-07 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Late Lumen Loss | 9 months post index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Windecker, MD, Principal Investigator — University Hospital (Inselspital) / Bern / Switzerland; Thierry Lefèvre, MD, Principal Investigator — Institute Hospitalier Jaques Cartier / Massy / France
Locations (24):
- Klinikum Wels-Grieskirchen, Wels, Upper Austria, Austria
- France (3):
  - Hospital Prive Jacques Cartier Massy, Massy
  - CHU - Hospital Arnaud de Villeneuve, Montpellier
  - Polyclinique les Fleurs Ollioules, Ollioules
- Germany (9):
  - Heart Centre Bad Krozingen, Bad Krozingen
  - Heart- and Diabetescentre NRW, Bad Oeyenhausen
  - Segeberger Kliniken GmbH, Bad Segeberg
  - Charité Campus Mitte, Berlin
  - Charité Campus Benjamin Franklin, Berlin
  - Universityhospital Lübeck, Lübeck
  - Städtische Kliniken Neuss, Lukaskrankenhaus GmbH, Neuss
  - Klinikum Nuernberg Sued, Nuremberg
  - Universityhospital Rostock, Rostock
- Heart centre Semmelweis University, Budapest, Hungary
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- OLVG (Onze Lieve Vrouwe Gasthuis), Amsterdam, Netherlands
- Spain (3):
  - Hospital Clínico y Provincial de Barcelona, Barcelona
  - Hospital Universitario Puerta de Hierro de Majadahonda, Madrid
  - Hospital Universitario Virgen de la Macarena, Seville
- Switzerland (5):
  - Cardiocentro Ticino, Lugano, Canton Ticino
  - University Hospital of Bern (Inselspital), Bern
  - University Hospital of Fribourg, Fribourg
  - University Hospital of Geneva, Geneva
  - Cantone Hospital of Lucerne, Lucerne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lefevre T, Haude M, Neumann FJ, Stangl K, Skurk C, Slagboom T, Sabate M, Goicolea J, Barragan P, Cook S, Macia JC, Windecker S. Comparison of a Novel Biodegradable Polymer Sirolimus-Eluting Stent With a Durable Polymer Everolimus-Eluting Stent: 5-Year Outcomes of the Randomized BIOFLOW-II Trial. JACC Cardiovasc Interv. 2018 May 28;11(10):995-1002. doi: 10.1016/j.jcin.2018.04.014. PMID 29798778
- [Derived] Mankerious N, Toelg R, Abdelghani M, Garcia-Garcia HM, Farhan S, Allali A, Windecker S, Lefevre T, Saito S, Kandzari DE, Waksman R, Richardt G, Hemetsberger R. Impact of coronary artery tortuosity on outcomes following stenting with newer-generation drug-eluting stents. An analysis of the randomized BIOFLOW trials. Rev Esp Cardiol (Engl Ed). 2025 Aug;78(8):682-691. doi: 10.1016/j.rec.2024.12.009. Epub 2025 Jan 4. English, Spanish. PMID 39761745
- [Derived] Hemetsberger R, Mankerious N, Toelg R, Abdelghani M, Farhan S, Garcia-Garica HM, Allali A, Windecker S, Lefevre T, Saito S, Kandzari D, Waksman R, Richardt G. Patients with higher-atherothrombotic risk vs. lower-atherothrombotic risk undergoing coronary intervention with newer-generation drug-eluting stents: an analysis from the randomized BIOFLOW trials. Clin Res Cardiol. 2023 Sep;112(9):1278-1287. doi: 10.1007/s00392-023-02205-4. Epub 2023 Apr 16. PMID 37062047
- [Derived] Hemetsberger R, Abdelghani M, Toelg R, Garcia-Garcia HM, Farhan S, Mankerious N, Elbasha K, Allali A, Windecker S, Lefevre T, Saito S, Kandzari D, Waksman R, Richardt G. Complex vs. non-complex percutaneous coronary intervention with newer-generation drug-eluting stents: an analysis from the randomized BIOFLOW trials. Clin Res Cardiol. 2022 Jul;111(7):795-805. doi: 10.1007/s00392-022-01994-4. Epub 2022 Feb 25. PMID 35212802
- [Derived] Hemetsberger R, Abdelghani M, Toelg R, Mankerious N, Allali A, Garcia-Garcia HM, Windecker S, Lefevre T, Saito S, Slagboom T, Kandzari D, Koolen J, Waksman R, Richardt G. Impact of Coronary Calcification on Clinical Outcomes After Implantation of Newer-Generation Drug-Eluting Stents. J Am Heart Assoc. 2021 Jun 15;10(12):e019815. doi: 10.1161/JAHA.120.019815. Epub 2021 May 29. PMID 34056911
- [Derived] Dan K, Garcia-Garcia HM, Kolm P, Windecker S, Saito S, Kandzari DE, Waksman R. Comparison of Ultrathin, Bioresorbable-Polymer Sirolimus-Eluting Stents and Thin, Durable-Polymer Everolimus-Eluting Stents in Calcified or Small Vessel Lesions. Circ Cardiovasc Interv. 2020 Sep;13(9):e009189. doi: 10.1161/CIRCINTERVENTIONS.120.009189. Epub 2020 Sep 8. PMID 32895004
- [Derived] Toelg R, Slagboom T, Waltenberger J, Lefevre T, Saito S, Kandzari DE, Koolen J, Richardt G. Individual patient data analysis of the BIOFLOW study program comparing safety and efficacy of a bioresorbable polymer sirolimus eluting stent to a durable polymer everolimus eluting stent. Catheter Cardiovasc Interv. 2021 Nov 1;98(5):848-856. doi: 10.1002/ccd.29254. Epub 2020 Sep 5. PMID 32890442
- [Derived] Windecker S, Haude M, Neumann FJ, Stangl K, Witzenbichler B, Slagboom T, Sabate M, Goicolea J, Barragan P, Cook S, Piot C, Richardt G, Merkely B, Schneider H, Bilger J, Erne P, Waksman R, Zaugg S, Juni P, Lefevre T. Comparison of a novel biodegradable polymer sirolimus-eluting stent with a durable polymer everolimus-eluting stent: results of the randomized BIOFLOW-II trial. Circ Cardiovasc Interv. 2015 Feb;8(2):e001441. doi: 10.1161/CIRCINTERVENTIONS.114.001441. PMID 25634905